CLINICAL TRIAL: NCT02696434
Title: A Phase 3, Randomized, Double-blind, Placebo-controlled, Parallel Group Study to Evaluate the Safety, Tolerability, and Efficacy of Naltrexone for Use in Conjunction With Buprenorphine in Adults With Opioid Use Disorder Transitioning From Buprenorphine Maintenance Prior to First Dose of VIVITROL
Brief Title: Evaluating Naltrexone for Use in Conjunction With Buprenorphine in Adults With Opioid Use Disorder Transitioning From Buprenorphine Maintenance Prior to First Dose of VIVITROL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alkermes, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ALK6428-A302
Record Dates: First submitted 2016-02-26; First posted 2016-03-02 (Estimated); Results first posted 2019-02-12 (Actual); Last update posted 2019-02-12 (Actual); Status verified 2019-01

CONDITIONS: Opioid Use Disorder
Keywords: naltrexone; VIVITROL; buprenorphine; opioid; addiction
MeSH Terms: conditions — Opioid-Related Disorders; Behavior, Addictive | interventions — Naltrexone; Buprenorphine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- PBO NTX + BUP (Active Comparator): Placebo naltrexone + buprenorphine
  Interventions: Drug: Placebo; Drug: Buprenorphine
- NTX + BUP (Experimental): Naltrexone + buprenorphine
  Interventions: Drug: Naltrexone; Drug: Buprenorphine

INTERVENTIONS:
Drug: Naltrexone — daily dosing
  Arms: NTX + BUP
Drug: Placebo — daily dosing
  Arms: PBO NTX + BUP
Drug: Buprenorphine — daily dosing

SUMMARY:
This study will evaluate the efficacy, safety, and tolerability of oral naltrexone used in conjunction with buprenorphine in adults with Opioid Use Disorder transitioning from buprenorphine maintenance prior to the first dose of VIVITROL.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide informed consent
* Willing and able to provide government-issued identification
* Has a Body Mass Index (BMI) of 18.0-40.0 kg/m^2
* Has a history of opioid use disorder diagnosis for at least 6 months
* Has a history of prescribed buprenorphine (or buprenorphine/naloxone) maintenance for the prior 3 or more consecutive months and is currently buprenorphine-maintained
* Must be voluntarily seeking treatment for opioid use disorder and be motivated to receive antagonist therapy
* Willing to abide by the contraception requirements for the duration of the study
* Additional criteria may apply

Exclusion Criteria:

* Is pregnant, planning to become pregnant or breastfeeding during the study
* Has a positive urine drug screen for opiates or oxycodone at screening
* Has used methadone within 30 days prior to study Day -5
* Has used naltrexone (oral or VIVITROL) within the 90 days prior to Day -5
* Has a history of seizures or has received anticonvulsant therapy within the past 5 years for treatment of seizures (use of anticonvulsant during the past detoxification is not exclusionary)
* Has a condition, disease state, or previous medical history that would preclude safe participation in the study or affect the ability to adhere to the protocol visit schedule, requirements, or assessments
* Has a current diagnosis of schizoaffective disorder, bipolar disorder, or untreated and unstable major depressive disorder
* Is currently physiologically dependent on any psychoactive substance (except opioids, caffeine, or nicotine) requiring medical intervention for detoxification
* Has a history of hypersensitivity or adverse reaction to buprenorphine, naltrexone, VIVITROL, or naloxone
* Additional criteria may apply

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 101 (Actual)
Dates: Start 2016-04; Primary Completion 2017-11 (Actual); Study Completion 2017-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria A. Sullivan, MD, PhD, Study Director — Alkermes, Inc.
Locations (9):
- United States (9):
  - Segal Institute for Clinical Research, Lauderhill, Florida
  - Research Centers of America, LLC, Oakland Park, Florida
  - Neuroscience Research Institute, Inc., Winfield, Illinois
  - John Hopkins School of Medicine, Baltimore, Maryland
  - Hassman Research Institute, Berlin, New Jersey
  - New York State Psychiatric Institute, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - University of Pennsylvania Treatment Research Center, Philadelphia, Pennsylvania
  - Western Psychiatric Institute and Clinic of University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mannelli P, Douaihy AB, Akerman SC, Legedza A, Fratantonio J, Zavod A, Sullivan MA. Characteristics and treatment preferences of individuals with opioid use disorder seeking to transition from buprenorphine to extended-release naltrexone in a residential setting. Am J Addict. 2022 Mar;31(2):142-147. doi: 10.1111/ajad.13264. Epub 2022 Feb 9. PMID 35137481
- [Derived] Mannelli P, Douaihy AB, Zavod A, Legedza A, Akerman SC, Sullivan MA. Patterns of withdrawal in patients with opioid use disorder (OUD) transitioning from untreated OUD or buprenorphine treatment to extended-release naltrexone. Am J Drug Alcohol Abuse. 2021 Nov 2;47(6):753-759. doi: 10.1080/00952990.2021.1969659. Epub 2021 Nov 9. PMID 34752714
- [Derived] Kosten T, Aharonovich E, Nangia N, Zavod A, Akerman SC, Lopez-Bresnahan M, Sullivan MA. Cognitive performance of patients with opioid use disorder transitioned to extended-release injectable naltrexone from buprenorphine: Post hoc analysis of exploratory results of a phase 3 randomized controlled trial. Addict Behav. 2020 Dec;111:106538. doi: 10.1016/j.addbeh.2020.106538. Epub 2020 Jul 3. PMID 32777606

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There is one subject who was randomized to the naltrexone + buprenorphine treatment arm, but mistakenly received placebo naltrexone + buprenorphine treatment. This subject is categorized in the PBO NTX+BUP arm in the participant flow and safety analyses, but in the efficacy analyses the subject is categorized as NTX+BUP.
Period: Overall Study
Arm/Group | NTX + BUP | PBO NTX + BUP
Started | 50 | 51
Completed | 28 | 33
Not Completed | 22 | 18
Not completed — Adverse Event | 3 | 1
Not completed — Lost to Follow-up | 5 | 4
Not completed — Withdrawal by Subject | 14 | 12
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NTX + BUP | PBO NTX + BUP | Total
Number analyzed (Participants) | 50 | 51 | 101
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.3 (9.41) | 34.8 (7.58) | 35.6 (8.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 16 | 30
  Male | 36 | 35 | 71
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 5
  Not Hispanic or Latino | 48 | 48 | 96
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 4 | 3 | 7
  White | 46 | 47 | 93
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 50 | 51 | 101

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects Who Receive and Tolerate a VIVITROL Injection on Day 8
Description: Demonstrated by mild opioid withdrawal symptoms (Clinical Opiate Withdrawal Scale [COWS] </=12 or Subjective Opiate Withdrawal Scale [SOWS] </=10) following VIVITROL administration. The COWS is a clinician-rated questionnaire designed to measure 11 common opioid withdrawal signs or symptoms. The summed score provides information about the level of physical dependence on opioids. The range of COWS scores is 0-4 (none to minimal); 5-12 (mild); 13-24 (moderate); 25-36 (moderately severe); and 37-48 (severe withdrawal). The SOWS is a 16-item self-report questionnaire designed to measure the severity of opioid withdrawal symptoms. The subject rates the intensity of symptoms using a 5-point scale. The range of SOWS scores is 1-10 (mild); 11-20 (moderate); and 21-30 (severe).
Time Frame: 8 days
Population: There is one subject who was randomized to the naltrexone + buprenorphine treatment arm, but mistakenly received placebo naltrexone + buprenorphine treatment. This subject is categorized in the PBO NTX+BUP arm in the participant flow and safety analyses, but in the efficacy analyses the subject is categorized as NTX+BUP.
Measure: Count of Participants; unit: Participants
Arm/Group | NTX + BUP | PBO NTX + BUP
Number analyzed (Participants) | 51 | 50
Participants | 35 | 38
Statistical Analysis 1: Comparison: NTX + BUP vs PBO NTX + BUP; Test type: Superiority; p = 0.407, Regression, Logistic; Odds Ratio (OR) = 0.68, 95% CI 2-sided [0.28 to 1.68]

2. Secondary Outcome: Proportion of Days With COWS Peak Score </=12 During the Treatment Period Prior to the VIVITROL Injection
Description: The Clinical Opiate Withdrawal Scale (COWS) is a clinician-rated questionnaire designed to measure 11 common opioid withdrawal signs or symptoms. The summed score provides information about the level of physical dependence on opioids. The range of COWS scores is 0-4 (none to minimal); 5-12 (mild); 13-24 (moderate); 25-36 (moderately severe); and 37-48 (severe withdrawal).
Time Frame: 1 week
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | NTX + BUP | PBO NTX + BUP
Number analyzed (Participants) | 51 | 50
Days | 5.8 (1.61) | 6.3 (1.36)

3. Secondary Outcome: Proportion of Post-VIVITROL Days (Days 9-11) in Which Subjects in Each Group Demonstrate Mild Opioid Withdrawal
Description: COWS score </=12; The Clinical Opiate Withdrawal Scale (COWS) is a clinician-rated questionnaire designed to measure 11 common opioid withdrawal signs or symptoms. The summed score provides information about the level of physical dependence on opioids. The range of COWS scores is 0-4 (none to minimal); 5-12 (mild); 13-24 (moderate); 25-36 (moderately severe); and 37-48 (severe withdrawal).
Time Frame: Days 9-11
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | NTX + BUP | PBO NTX + BUP
Number analyzed (Participants) | 51 | 50
Days | 2.4 (0.87) | 2.6 (0.81)

4. Secondary Outcome: Mean Peak COWS Scores During the Treatment Period (Days 1/1a-7)
Description: as for outcome 2
Time Frame: Up to 7 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NTX + BUP | PBO NTX + BUP
Number analyzed (Participants) | 51 | 50
score on a scale | 6.0 (3.71) | 5.0 (2.78)

5. Secondary Outcome: Area Under the Curve (AUC) for COWS Scores During the Treatment Period and VIVITROL Induction and Post-VIVITROL Observation Period
Description: The Clinical Opiate Withdrawal Scale (COWS) is a clinician-rated questionnaire designed to measure 11 common opioid withdrawal signs or symptoms. The summed score provides information about the level of physical dependence on opioids. The range of COWS scores is 0-4 (none to minimal); 5-12 (mild); 13-24 (moderate); 25-36 (moderately severe); and 37-48 (severe withdrawal). The daily AUC COWS score is derived based on the actual time (unit in minutes) COWS administered on each day by using the linear trapezoidal rule, and then divided by the COWS administration duration (last COWS administration time minus first COWS administration time) for that day. The normalized AUC COWS score is the summation of daily AUC COWS score during the relevant period divided by the number of days with daily AUC COWS score.
Time Frame: The COWS was administered 4-6 times per day during the Treatment Period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NTX + BUP | PBO NTX + BUP
Number analyzed (Participants) | 51 | 50
score on a scale | 4.5 (3.11) | 3.9 (2.29)

6. Secondary Outcome: Mean Score for "Desire for Opioids" Visual Analog Scale (VAS) During the Treatment Period and VIVITROL Induction and Post-VIVITROL Observation Period
Description: The Desire for Opioids VAS uses a 100-mm, horizontal linear scale, with 0 anchored on the left representing "no desire for opioids" and 100 anchored on the right representing "strongest imaginable desire for opioids."
Time Frame: Up to 11 days
Population: All randomized subjects who received at least 1 dose of study drug and provided at least 1 post-baseline measureable VAS assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NTX + BUP | PBO NTX + BUP
Number analyzed (Participants) | 45 | 46
score on a scale | 6.3 (12.62) | 8.3 (14.43)

7. Secondary Outcome: Incidence of Adverse Events (AEs)
Description: Number and percentage of subjects who experienced AEs.
Time Frame: Up to 42 days
Population: There is one subject who was randomized to the naltrexone + buprenorphine treatment arm, but mistakenly received placebo naltrexone + buprenorphine treatment. All the efficacy analyses are summarized by the planned treatment assignment, and all the safety analyses are summarized by actual treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | NTX + BUP | PBO NTX + BUP
Number analyzed (Participants) | 50 | 51
Participants | 38 | 37

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over a period of 42 days
Arm/Group | NTX + BUP | PBO NTX + BUP
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/51
Serious Adverse Events (participants affected / at risk) | 0/50 | 1/51
Other Adverse Events (participants affected / at risk) | 36/50 | 34/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NTX + BUP (N=50) | PBO NTX + BUP (N=51)
Suicidal Ideation (Psychiatric disorders) | 0 (0) | 1 (1)
Psychotic Disorder (Psychiatric disorders) | 0 (0) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NTX + BUP (N=50) | PBO NTX + BUP (N=51)
Anxiety (Psychiatric disorders) | 15 (15) | 15 (15)
Insomnia (Psychiatric disorders) | 13 (14) | 13 (13)
Restlessness (Psychiatric disorders) | 4 (4) | 5 (5)
Drug Withdrawal Syndrome (Psychiatric disorders) | 3 (5) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 16 (16) | 9 (9)
Nausea (Gastrointestinal disorders) | 9 (10) | 5 (5)
Abdominal Pain Upper (Gastrointestinal disorders) | 7 (7) | 6 (6)
Constipation (Gastrointestinal disorders) | 3 (3) | 6 (6)
Dyspepsia (Gastrointestinal disorders) | 3 (3) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 10 (10) | 6 (6)
Back Pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Headache (Nervous system disorders) | 5 (7) | 3 (3)
Restless Legs Syndrome (Nervous system disorders) | 3 (4) | 0 (0)
Pain (General disorders) | 3 (3) | 4 (4)
Fatigue (General disorders) | 2 (2) | 3 (3)
Hypotension (Vascular disorders) | 4 (4) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Should an Investigator desire to disclose study results, Sponsor will review the results disclosure prior to public release and can embargo the disclosure for a period of at least 60 days. Revisions to the disclosure will be negotiated in good faith. For a multicenter study the Investigators agree to publish/publicly present the results together with the other sites for the 12 month period after study results are available unless Sponsor grants written permission in advance.

DOCUMENTS (2):
  • Study Protocol (2017-06-14): https://cdn.clinicaltrials.gov/large-docs/34/NCT02696434/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-29): https://cdn.clinicaltrials.gov/large-docs/34/NCT02696434/SAP_001.pdf